CLINICAL TRIAL: NCT04143867
Title: A Feasibility Efficacy and Safety Study of the Nolix Vaginal Device for the Temporary Management of Stress Urinary Incontinence in Women
Brief Title: The Nolix Feasibility Efficacy and Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynamics LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NLX-002
Record Dates: First submitted 2019-10-22; First posted 2019-10-29 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: A prospective, one-arm study with subjects serving as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nolix Device (Experimental): Comparing use of device to non-treatment (pads only) phase
  Interventions: Device: Nolix Device

INTERVENTIONS:
Device: Nolix Device — For temporary management of SUI

SUMMARY:
This study is an open label, prospective, feasibility study with the Nolix device used for temporary treatment of Stress Urinary Incontinence (SUI) in subjects, serving as their own controls.

DETAILED DESCRIPTION:
This is an open label, prospective, feasibility study with the Nolix device used in subjects with SUI, serving as their own controls. The objective of this study is to evaluate the effectiveness (both objective and subjective) and safety of the Nolix device when used for the temporary management of SUI in women. In addition, the study is aimed to evaluate changes in the quality of life (QoL) and comfort during use of the Nolix device. The primary effectiveness endpoint is the percent change in the mean Pad Weight Gain (%PWG) between the device (during the last 7 days of the 14-days Nolix use period) and control periods , with the success criterion defined as at least >-50% of the mean %PWG change during the last 7 days of the treatment phase as compared to the control phase. Additional effectiveness endpoints include the number of self-reported SUI episodes per week, the percentage of subjects who experience a greater than -50% change in the number of self-reported daily incontinence episodes, as well as the changes in the QoL, leak scores and overall satisfaction levels. The safety of the Nolix device is also evaluated by assessing the adverse events, including the results of urinalysis, vaginal swab, and vaginal examination.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 22 and above.
* Suffering from Stress Urinary Incontinence.
* Women who can understand the nature of the study, are physically able to perform all required tasks and consent to it by signing a written Informed Consent Form prior to participation in the study.

Exclusion Criteria:

* Age ≤ 21 years.
* Pregnant or planning to become pregnant during the study.
* Vaginal birth or Cesarean section for the last 3 months prior to entering the study.
* Severely atrophic vagina.
* A history of Toxic Shock Syndrome (TSS).
* Active urinary tract or vaginal infection.
* Patients prone to recurrent vaginal or urinary tract infections (i.e. more than 3 times in the past year).
* Has experienced unusual or unexpected vaginal bleeding within the last 6 months.
* Vaginal surgery within the last 3 months prior to entering the study.
* Has experienced difficulties with the use of intra-vaginal devices, including tampons.
* Presence of any condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Average daily PWG as measured in the baseline pad period is less than 4 grams /12 hours.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Mean pad weight gain (PWG) change of >50% when comparing the PWG control phase as compared to the Nolix device phase. | 21 days
  The primary effectiveness endpoint is the percent change in the mean Pad Weight Gain (%PWG) between the device (during the last 7 days of the 14-days Nolix use period) and control periods , with the success criterion defined as at least >50% of the mean %PWG reduction during the last 7 days of the treatment phase as compared to the control phase.
Device-related adverse events | 21 days
  Discomfort / pain, vaginal irritation or itching, vaginal spotting, vaginal or urinary tract infections

SECONDARY OUTCOMES:
Change in number of self-reported incontinence episodes. | 21 days
  Change in number of self-reported incontinence episodes per week from the control period to the Nolix device use period.
More than 50% reduction in the number of self-reported daily incontinence episodes. | 21 days
  Percentage of subjects who experience a greater than 50% reduction in the number of self-reported daily incontinence episodes from the baseline period to the Nolix device use period.
Changes in Quality of Life (QoL). | 21 days
  The QoL Questionnaire (measured on a 0-100 scale) will be performed at baseline and after the device-use period and refer to areas which may have been influenced or changed by accidental urine loss and/or prolapse. A lower score is considered less impact to quality of life and a higher score reflects more impact to quality of life. In the same manner, a reduction in scores from baseline reflects improved quality of life.
Changes in Leak Score. | 21 days
  Changes in Leak Score from the baseline period to the Nolix device use period, as measured using the Leak Score Questionnaire. The Leak Score Questionnaire will be performed (on a 0-3 scale) to evaluate the subjective perception of incontinence during eight effort demanding activities: coughing, laughing, sneezing, jumping, lifting heavy objects, walking, running, and going to the gym.
PWG measured continuously. | 21 days
  PWG measured continuously (as opposed to responder analysis), using the same definition of PWG as described above, without transformation to percent.
Comfort during Nolix device use. | 21 days
  Comfort during Nolix device use will be measured through the Satisfaction Questionnaire, using a 10-point scale (where 1 is the most negative response and 10 the most positive, during the use of the device).
Overall perception of improvement. | 21 days
  Overall perception of improvement following the use of the Nolix device, as measured using the Patient Global Impression of Improvement (PGI-I) Scale, measured on a 7-point scale (where 1 is the most positive response and 7 the most negative response).
Overall satisfaction: Patient Satisfaction Question (PSQ) | 21 days
  Overall satisfaction with the use of the Nolix device, as measured using the Patient Satisfaction Question (PSQ),selecting one of the following answers: 'Completely'; 'Somewhat'; or 'Not at all'.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Fridman, Dr., Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
All personal data gathered in this trial will be treated in strictest confidence by investigators, monitors, sponsor's personnel and independent ethics committee.